CLINICAL TRIAL: NCT04804813
Title: Drug Use Surveillance for Cabometyx Tablets "Renal Cell Carcinoma"
Brief Title: Survey of Cabozantinib Used To Treat People With Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Cabozantinib-5001; jRCT2031210003 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cabozantinib 60 mg: Cabozantinib 60 milligrams (mg) tablet, orally, once daily for up to 26 weeks. Participants received interventions as part of routine medical care.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib tablets
  Other Names: Cabometyx tablets

SUMMARY:
This study is a survey in Japan of Cabozantinib tablets used to treat people with a type of kidney cancer called renal cell carcinoma. The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects from Cabozantinib. During the study, participants with renal cell carcinoma will take Cabozantinib tablets according to their clinic's standard practice. The study doctors will check for side effects from Cabozantinib for 26 weeks.

DETAILED DESCRIPTION:
The drug being tested in this study is called cabozantinib tablets. This tablet is being tested to treat people who have radically unresectable or metastatic renal cell carcinoma.

This study is an observational (non-interventional) study and will look at occurrence of adverse drug reactions (or adverse events) of cabozantinib tablets in the routine clinical setting. The planned number of observed patients will be approximately 300.

This multi-center observational trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

Patients with radically unresectable or metastatic renal cell carcinoma who do not meet the following exclusion criterion are eligible.

Exclusion Criteria:

A patient who has a history of hypersensitivity to any component of cabozantinib.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with radically unresectable or metastatic renal cell carcinoma as part of routine medical care
Sampling Method: Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/606d5f0c620b3b001e9dbb51

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 102 investigative sites in Japan, from 29 March 2021 to 25 July 2024.
Pre-assignment Details: Participants with renal cell carcinoma who received Cabozantinib were enrolled. Participants received Cabozantinib as part of a routine medical care.
Groups:
- Cabozantinib Monotherapy: Participants with renal cell carcinoma who received Cabozantinib 60 milligrams (mg) tablet, orally, once daily for up to 26 weeks as part of routine medical care.
- Cabozantinib + Nivolumab Combination Therapy: Participants with renal cell carcinoma who received Cabozantinib 40 milligrams (mg) tablet, orally, once daily, and Nivolumab intravenous infusion as part of routine medical care.
Period: Overall Study
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Started | 325 | 63
Completed | 322 | 63
Not Completed | 3 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy | Total
Number analyzed (Participants) | 322 | 63 | 385
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (11.34) | 68.7 (11.55) | 68.7 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 17 | 115
  Male | 224 | 46 | 270
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAE)
Description: An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. An SAE is any event that results in: death; life-threatening; requires inpatient hospitalization or results in prolongation of existing hospitalization; persistent or significant disability/incapacity; a congenital anomaly/birth defect or a medically important event.
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Participants
  Adverse Events | 216 | 46
  Serious Adverse Events | 73 | 28

2. Primary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: Severity grade is defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Participants | 103 | 29

3. Primary Outcome: Percentage of Adverse Events Leading to Dose Changes of Cabozantinib
Description: An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Number; unit: Percent of Adverse Events
Units Other Than Participants: Count of Adverse Events
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Number analyzed (Count of Adverse Events) | 425 | 92
Percent of Adverse Events | 72.0 | 64.1

4. Primary Outcome: Number of Participants With Adverse Drug Reactions and Serious Adverse Drug Reactions
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any event that results in: death; life-threatening; requires inpatient hospitalisation or results in prolongation of existing hospitalisation; persistent or significant disability/incapacity; a congenital anomaly/birth defect or a medically important event. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Participants
  Adverse Drug Reactions | 193 | 41
  Serious Adverse Drug Reactions | 49 | 18

5. Primary Outcome: Number of Participants With Grade 3 or Higher Adverse Drug Reactions
Description: as for outcome 2
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Participants | 80 | 24

6. Primary Outcome: Percentage of Adverse Drug Reactions Leading to Dose Changes of Cabozantinib
Description: as for outcome 4
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Number; unit: Percent of Adverse Drug Reactions
Units Other Than Participants: Count of Adverse Drug Reactions
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Number analyzed (Count of Adverse Drug Reactions) | 373 | 70
Percent of Adverse Drug Reactions | 72.1 | 74.3

7. Primary Outcome: Number of Participants With Adverse Drug Reaction and Serious Adverse Drug Reactions of Hepatic Failure and Hepatic Dysfunction
Description: as for outcome 4
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Participants
  Adverse Drug Reaction of Hepatic Failure and Hepatic Dysfunction | 52 | 16
  Serious Adverse Drug Reactions of Hepatic Failure and Hepatic Dysfunction | 2 | 4

8. Primary Outcome: Number of Participants With Grade 3 or Higher Adverse Drug Reactions of Hepatic Failure and Hepatic Dysfunction
Description: as for outcome 2
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Participants | 8 | 7

9. Primary Outcome: Percentage of Adverse Drug Reactions of Hepatic Failure and Hepatic Dysfunction Leading to Dose Changes of Cabozantinib
Description: as for outcome 4
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Number; unit: Percent of Adverse Drug Reactions
Units Other Than Participants: Count of Adverse Drug Reactions
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Number analyzed (Count of Adverse Drug Reactions) | 61 | 19
Percent of Adverse Drug Reactions | 77.0 | 78.9

10. Primary Outcome: Number of Participants With Adverse Drug Reaction and Serious Adverse Drug Reactions of Pancreatitis
Description: as for outcome 4
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Participants
  Adverse Drug Reaction of Pancreatitis | 9 | 3
  Serious Adverse Drug Reactions of Pancreatitis | 4 | 1

11. Primary Outcome: Number of Participants With Grade 3 or Higher Adverse Drug Reactions of Pancreatitis
Description: as for outcome 2
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Participants | 2 | 3

12. Primary Outcome: Percentage of Adverse Drug Reactions of Pancreatitis Leading to Dose Changes of Cabozantinib
Description: as for outcome 4
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Number; unit: Percent of Adverse Drug Reactions
Units Other Than Participants: Count of Adverse Drug Reactions
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Number analyzed (Count of Adverse Drug Reactions) | 10 | 4
Percent of Adverse Drug Reactions | 50.0 | 100.0

13. Secondary Outcome: Percentage of Participants Who Achieve or Maintain Any Best Response
Description: Best response was assessed with reference to the excerpts from Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Best response was defined as the level of best response in assessment with complete response (CR), partial response (PR) during the observational period.
Time Frame: Up to 26 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
Number analyzed (Participants) | 322 | 63
Participants | 106 | 26

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Cabozantinib Monotherapy | Cabozantinib + Nivolumab Combination Therapy
All-Cause Mortality (participants affected / at risk) | 15/322 | 5/63
Serious Adverse Events (participants affected / at risk) | 73/322 | 28/63
Other Adverse Events (participants affected / at risk) | 165/322 | 24/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib Monotherapy (N=322) | Cabozantinib + Nivolumab Combination Therapy (N=63)
Peritonitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pneumonia aspiration (Infections and infestations) | 2 | 0
Retroperitoneal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Subperiosteal abscess (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 2
Metastases to heart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 2
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 8 | 3
Thyroiditis (Endocrine disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Vitreoretinal traction syndrome (Eye disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 4
Liver disorder (Hepatobiliary disorders) | 0 | 1
Gallbladder enlargement (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Death (General disorders) | 1 | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Malaise (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 1 | 0
Mucosal disorder (General disorders) | 1 | 0
Amylase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib Monotherapy (N=322) | Cabozantinib + Nivolumab Combination Therapy (N=63)
Decreased appetite (Metabolism and nutrition disorders) | 17 | 2
Hypertension (Vascular disorders) | 28 | 4
Diarrhoea (Gastrointestinal disorders) | 35 | 4
Stomatitis (Gastrointestinal disorders) | 17 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 28 | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 40 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT04804813/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT04804813/SAP_001.pdf